CLINICAL TRIAL: NCT01390428
Title: An Open-label, 3-Part, Multiple Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of Grazoprevir (MK-5172)
Brief Title: Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of Grazoprevir (MK-5172-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-013
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1-Mild Hepatic Impairment (HI) (Experimental): Participants with mild hepatic impairment will receive 200 mg of Grazoprevir once a day for 10 consecutive days during Part 1 of the study.
  Interventions: Drug: Grazoprevir
- Part 1-Healthy Matched to Mild HI (Experimental): Healthy participants will receive 200 mg of Grazoprevir once a day for 10 consecutive days during Part 1 of the study.
  Interventions: Drug: Grazoprevir
- Part 2-Moderate HI (Experimental): Participants with moderate hepatic impairment will receive 100 mg of Grazoprevir once a day for 10 consecutive days during Part 2 of the study.
  Interventions: Drug: Grazoprevir
- Part 2-Healthy Matched to Moderate HI (Experimental): Healthy participants will receive 100 mg of Grazoprevir once a day for 10 consecutive days during Part 2 of the study.
  Interventions: Drug: Grazoprevir
- Part 3-Severe HI (Experimental): Participants with severe hepatic impairment will receive 50 mg of Grazoprevir once a day for 10 consecutive days during Part 3 of the study.
  Interventions: Drug: Grazoprevir
- Part 3-Healthy Matched to Severe HI (Experimental): Healthy participants will receive 50 mg of Grazoprevir once a day for 10 consecutive days during Part 3 of the study.
  Interventions: Drug: Grazoprevir

INTERVENTIONS:
Drug: Grazoprevir — Part 1: oral morning dose of 200 mg daily for 10 days Part 2: oral morning dose of 100 mg daily for 10 days Part 3: oral morning dose of 50 mg daily for 10 days

SUMMARY:
This study will compare the pharmacokinetics (PK) of grazoprevir (MK-5172) when administered to participants with mild, moderate or severe hepatic insufficiency (assessed by the criteria of the Child-Pugh's scale) with the PK of grazoprevir when administered to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be of non-childbearing potential or willing to use at least 2 acceptable methods of contraception from enrollment to 2 weeks after the last dose of study drug
* No clinically significant abnormality on electrocardiogram

Hepatic Insufficiency Participants Only:

* Other than hepatic insufficiency with features of cirrhosis, is otherwise in good health based on medical history, physical examination, vital signs, and laboratory safety tests
* Chronic (>6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology
* Score on the Child-Pugh scale must range from 5 to 6 (mild hepatic insufficiency) to from 7 to 9 (moderate hepatic insufficiency) to from 10 to 15 (severe hepatic insufficiency)

Matched Healthy Participants Only:

- In good health based on medical history, physical examination, vital signs, and laboratory safety tests

Exclusion Criteria:

* History of any illness that might confound the results of the study or poses an additional risk to the participant
* History of clinically significant endocrine, gastrointestinal (other than related to their hepatic impairment), cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Pregnancy
* Estimated creatinine clearance of ≤60 mL/min
* History of stroke, chronic seizures, or major neurological disorder
* History of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort, green tea, gingko, coenzyme Q, ginseng, echinacea, etc.) or nutritional supplements (e.g., garlic supplements), beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study, until the poststudy visit
* Participated in another investigational study within 4 weeks
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food

Hepatic Insufficiency Participants Only:

- Has a history of hepatitis C infection by serology, regardless of most recent viral load status.

Matched Healthy Participants Only:

* History of any chronic and/or active hepatic disease including elevations of serum transaminases, hepatitis, biliary tract disease, or a history of any significant gastrointestinal surgery.
* History of hepatitis C. Participants with a history of self-limited hepatitis A with complete resolution documented at least 6 months prior to entry will be eligible for inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2014-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Caro L, Wenning L, Guo Z, Fraser IP, Fandozzi C, Talaty J, Panebianco D, Ho M, Uemura N, Reitmann C, Angus P, Gane E, Marbury T, Smith WB, Iwamoto M, Butterton JR, Yeh WW. Effect of Hepatic Impairment on the Pharmacokinetics of Grazoprevir, a Hepatitis C Virus Protease Inhibitor. Antimicrob Agents Chemother. 2017 Nov 22;61(12):e00813-17. doi: 10.1128/AAC.00813-17. Print 2017 Dec. PMID 28947470

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1-Mild Hepatic Impairment (HI): Participants with mild HI received 200 mg of Grazoprevir once a day for 10 consecutive days during Part 1 of the study.
- Part 1-Healthy Matched to Mild HI: Healthy participants received 200 mg of Grazoprevir once a day for 10 consecutive days during Part 1 of the study.
- Part 2-Moderate HI: Participants with moderate HI received 100 mg of Grazoprevir once a day for 10 consecutive days during Part 2 of the study.
- Part 2-Healthy Matched to Moderate HI: Healthy participants received 100 mg of Grazoprevir once a day for 10 consecutive days during Part 2 of the study.
- Part 3-Severe HI: Participants with severe HI received 50 mg of Grazoprevir once a day for 10 consecutive days during Part 3 of the study.
- Part 3-Healthy Matched to Severe HI: Healthy participants received 50 mg of Grazoprevir once a day for 10 consecutive days during Part 3 of the study.
Period: Overall Study
Arm/Group | Part 1-Mild Hepatic Impairment (HI) | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Started | 8 | 8 | 9 | 9 | 8 | 8
Completed | 8 | 8 | 8 | 9 | 7 | 8
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Elective Surgery | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1-Mild HI: Participants with mild HI received 200 mg of Grazoprevir once a day for 10 consecutive days during Part 1 of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI | Total
Number analyzed (Participants) | 8 | 8 | 9 | 9 | 8 | 8 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (4.1) | 54.5 (5.8) | 53.3 (6.7) | 52.3 (6.8) | 52.1 (8.4) | 52.0 (9.9) | 53.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 0 | 3 | 3 | 12
  Male | 5 | 5 | 9 | 9 | 5 | 5 | 38

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time-curve From 0 to 24 Hours (AUC0-24) of Grazoprevir
Description: Blood samples were collected at pre-dose, and from 0.5 to 24 hours post-dose on Days 1 and 10 in order to determine the plasma AUC0-24 of Grazoprevir. Classification of HI based on the Child-Pugh scale, where a score of 5-6 = Mild HI; a score of 7-9 = Moderate HI; and a score of 10-15 = Severe HI.
Time Frame: Days 1 and 10 at the following timepoints: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: Participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
uM*hr
  Day 1 | 1.71 [1.10 to 2.65] | 1.42 [0.912 to 2.20] | 1.61 [0.791 to 3.29] | 0.321 [0.157 to 0.655] | 1.17 [0.541 to 2.55] | 0.0592 [0.0273 to 0.129]
  Day 10 | 6.20 [4.19 to 9.18] | 3.74 [2.53 to 5.54] | 4.21 [2.48 to 7.14] | 0.874 [0.515 to 1.48] | 3.00 [1.71 to 5.26] | 0.257 [0.146 to 0.451]
Statistical Analysis 1: Comparison: Part 1-Mild HI vs Part 1-Healthy Matched to Mild HI; Day 1; Test type: Superiority or Other; Geometric Least Squares Mean Ratio (GMR) = 1.21, 90% CI 2-sided [0.73 to 2.01] — Mild Hepatic Impairment (HI)/Healthy Matched to Mild HI
Statistical Analysis 2: Comparison: Part 1-Mild HI vs Part 1-Healthy Matched to Mild HI; Day 10; Test type: Superiority or Other; GMR = 1.66, 90% CI 2-sided [1.05 to 2.61] — Mild HI/Healthy Matched to Mild HI
Statistical Analysis 3: Comparison: Part 2-Moderate HI vs Part 2-Healthy Matched to Moderate HI; Day 1; Test type: Superiority or Other; GMR = 5.03, 90% CI 2-sided [2.19 to 11.56] — Moderate HI/Healthy Matched to Moderate HI
Statistical Analysis 4: Comparison: Part 2-Moderate HI vs Part 2-Healthy Matched to Moderate HI; Day 10; Test type: Superiority or Other; GMR = 4.82, 90% CI 2-sided [2.60 to 8.93] — Moderate HI/Healthy Matched to Moderate HI
Statistical Analysis 5: Comparison: Part 3-Severe HI vs Part 3-Healthy Matched to Severe HI; Day 1; Test type: Superiority or Other; GMR = 19.83, 90% CI 2-sided [8.11 to 48.51] — Severe HI/Healthy Matched to Severe HI
Statistical Analysis 6: Comparison: Part 3-Severe HI vs Part 3-Healthy Matched to Severe HI; Day 10; Test type: Superiority or Other; GMR = 11.68, 90% CI 2-sided [6.10 to 22.35] — Severe HI/Healthy Matched to Severe HI

2. Primary Outcome: Maximum Concentration (Cmax) of Grazoprevir
Description: Blood samples were collected at pre-dose, and from 0.5 to 24 hours post-dose on Days 1 and 10 in order to determine the plasma Cmax of Grazoprevir. Classification of HI based on the Child-Pugh scale, where a score of 5-6 = Mild HI; a score of 7-9 = Moderate HI; and a score of 10-15 = Severe HI.
Time Frame: Days 1 and 10 at the following timepoints: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: uM
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
uM
  Day 1 | 0.257 [0.121 to 0.545] | 0.305 [0.144 to 0.646] | 0.433 [0.184 to 1.07] | 0.0580 [0.0242 to 0.139] | 0.238 [0.107 to 0.531] | 0.0157 [0.00705 to 0.0350]
  Day 10 | 1.40 [0.903 to 2.17] | 1.02 [0.658 to 1.58] | 0.631 [0.334 to 1.19] | 0.106 [0.0559 to 0.199] | 0.396 [0.203 to 0.774] | 0.0304 [0.0156 to 0.0595]
Statistical Analysis 1: Comparison: Part 1-Mild HI vs Part 1-Healthy Matched to Mild HI; Day 1; Test type: Superiority or Other; GMR = 0.84, 90% CI 2-sided [0.35 to 2.01] — Mild HI/Healthy Matched to Mild HI
Statistical Analysis 2: Comparison: Part 1-Mild HI vs Part 1-Healthy Matched to Mild HI; Day 10; Test type: Superiority or Other; GMR = 1.37, 90% CI 2-sided [0.83 to 2.27] — Mild HI/Healthy Matched to Mild HI
Statistical Analysis 3: Comparison: Part 2-Moderate HI vs Part 2-Healthy Matched to Moderate HI; Day 1; Test type: Superiority or Other; GMR = 7.64, 90% CI 2-sided [2.74 to 21.27] — Moderate HI/Healthy Matched to Moderate HI
Statistical Analysis 4: Comparison: Part 2-Moderate HI vs Part 2-Healthy Matched to Moderate HI; Day 10; Test type: Superiority or Other; GMR = 5.98, 90% CI 2-sided [2.84 to 12.57] — Moderate HI/Healthy Matched to Moderate HI
Statistical Analysis 5: Comparison: Part 3-Severe HI vs Part 3-Healthy Matched to Severe HI; Day 1; Test type: Superiority or Other; GMR = 15.18, 90% CI 2-sided [6.02 to 38.25] — Severe HI/Healthy Matched to Severe HI
Statistical Analysis 6: Comparison: Part 3-Severe HI vs Part 3-Healthy Matched to Severe HI; Day 10; Test type: Superiority or Other; GMR = 13.01, 90% CI 2-sided [6.00 to 28.21] — Severe HI/Healthy Matched to Severe HI

3. Primary Outcome: Time to Peak Concentration (Tmax) of Grazoprevir
Description: Blood samples were collected at pre-dose, and from 0.5 to 24 hours post-dose on Days 1 and 10 in order to determine the plasma Tmax of Grazoprevir. Classification of HI based on the Child-Pugh scale, where a score of 5-6 = Mild HI; a score of 7-9 = Moderate HI; and a score of 10-15 = Severe HI.
Time Frame: Days 1 and 10 at the following timepoints: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr.
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
hr.
  Day 1 | 3.50 [1.00 to 12.00] | 2.50 [1.00 to 4.00] | 2.00 [1.50 to 4.00] | 1.75 [1.00 to 4.00] | 1.75 [1.00 to 3.00] | 1.50 [1.00 to 4.00]
  Day 10 | 3.00 [2.00 to 4.00] | 3.01 [1.5 to 4.00] | 3.00 [1.50 to 8.00] | 2.00 [1.00 to 6.00] | 1.75 [0.50 to 4.00] | 1.00 [0.50 to 3.00]

4. Primary Outcome: Concentrations 24 Hours Post-dose (C24) of Grazoprevir on Day 1 for Participants With Mild HI and Moderate HI and Healthy Matched to Mild HI and Moderate HI
Description: Blood samples were collected at 24 hours post-dose on Day 1 in order to determine the plasma C24 of Grazoprevir. Classification of HI based on the Child-Pugh scale, where a score of 5-6 = Mild HI; a score of 7-9 = Moderate HI; and a score of 10-15 = Severe HI.
Time Frame: Day 1 at 24 hours postdose
Population: Participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Participants with Severe HI and Matched Healthy to Severe HI are absent because they had a different Measure Type and Method of Dispersion
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 0
nM | 21.4 [18.2 to 25.2] | 11.5 [9.8 to 13.5] | 17.7 [8.73 to 35.8] | 5.90 [2.92 to 11.9] |  |
Statistical Analysis 1: Comparison: Part 1-Mild HI vs Part 1-Healthy Matched to Mild HI; Test type: Superiority or Other; GMR = 1.86, 90% CI 2-sided [1.54 to 2.24] — Mild HI/Healthy Matched to Mild HI
Statistical Analysis 2: Comparison: Part 2-Moderate HI vs Part 2-Healthy Matched to Moderate HI; Test type: Superiority or Other; GMR = 2.99, 90% CI 2-sided [1.31 to 6.82] — Moderate HI/Healthy Matched to Moderate HI

5. Primary Outcome: Concentrations 24 Hours Post-dose (C24) of Grazoprevir on Day 1 for Participants With Severe HI and Healthy Matched to Severe HI
Description: as for outcome 4
Time Frame: Day 1 at 24 hours postdose
Population: Participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Participants with Mild HI, Moderate HI and Healthy Matched to Mild HI or Moderate HI are absent because they had a different Measure Type and Method of Dispersion
Measure: Median (Full Range); unit: nM
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
nM |  |  |  |  | 15.6 [2.89 to 60.2] | 1.86 [0.00 to 3.32]

6. Primary Outcome: Concentrations 24 Hours Post-dose (C24) of Grazoprevir on Day 10
Description: Blood samples were collected at 24 hours post-dose on Day 10 in order to determine the plasma C24 of Grazoprevir. Classification of HI based on the Child-Pugh scale, where a score of 5-6 = Mild HI; a score of 7-9 = Moderate HI; and a score of 10-15 = Severe HI.
Time Frame: Days 10 at 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
nM | 32.6 [24.8 to 42.8] | 17.0 [12.9 to 22.3] | 48.9 [27.2 to 87.9] | 13.6 [7.60 to 24.5] | 55.0 [31.9 to 94.8] | 5.89 [3.42 to 10.2]
Statistical Analysis 1: Comparison: Part 1-Mild HI vs Part 1-Healthy Matched to Mild HI; Test type: Superiority or Other; GMR = 1.92, 90% CI 2-sided [1.40 to 2.63] — Mild HI/Healthy Matched to Mild HI
Statistical Analysis 2: Comparison: Part 2-Moderate HI vs Part 2-Healthy Matched to Moderate HI; Test type: Superiority or Other; GMR = 3.59, 90% CI 2-sided [1.81 to 7.11] — Moderate HI/Healthy Matched to Moderate HI
Statistical Analysis 3: Comparison: Part 3-Severe HI vs Part 3-Healthy Matched to Severe HI; Test type: Superiority or Other; GMR = 9.34, 90% CI 2-sided [4.98 to 17.51] — Severe HI/Healthy Matched to Severe HI

7. Primary Outcome: Apparent Terminal Half-life (t1/2) of Grazoprevir
Description: Blood samples were collected at pre-dose, and from 0.5 to 24 hours post-dose on Day 10 in order to determine the plasma t1/2 of Grazoprevir. Classification of HI based on the Child-Pugh scale, where a score of 5-6 = Mild HI; a score of 7-9 = Moderate HI; and a score of 10-15 = Severe HI.
Time Frame: Day 10 at the following timepoints: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
hr. | 54.24 (22.32) | 35.85 (47.15) | 39.59 (23.76) | 39.80 (17.34) | 42.00 (26.55) | 31.02 (41.99)

ADVERSE EVENTS:
Time Frame: 14 days after last dose (up to Day 24)
Arm/Group | Part 1-Mild HI | Part 1-Healthy Matched to Mild HI | Part 2-Moderate HI | Part 2-Healthy Matched to Moderate HI | Part 3-Severe HI | Part 3-Healthy Matched to Severe HI
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/9 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 5/8 | 4/9 | 4/9 | 4/8 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1-Mild HI (N=8) | Part 1-Healthy Matched to Mild HI (N=8) | Part 2-Moderate HI (N=9) | Part 2-Healthy Matched to Moderate HI (N=9) | Part 3-Severe HI (N=8) | Part 3-Healthy Matched to Severe HI (N=8)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1-Mild HI (N=8) | Part 1-Healthy Matched to Mild HI (N=8) | Part 2-Moderate HI (N=9) | Part 2-Healthy Matched to Moderate HI (N=9) | Part 3-Severe HI (N=8) | Part 3-Healthy Matched to Severe HI (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.